CLINICAL TRIAL: NCT06283316
Title: Systemic Treatments for Alopecia Areata Registry
Acronym: STA2R
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, DirkJan Hijnen, Principal Investigator, Erasmus Medical Center
Other Study IDs: 11347
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis; Hair Loss; Hair Diseases; Alopecia; Alopecia Drugs; Autoimmune Diseases
Keywords: Alopecia Areata; Alopecia Totalis; Alopecia Universalis; Systemic treatment; Registry
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia; Hair Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter prospective registry (STA2R) is conducted to assess systemic treatments for alopecia areata, focusing on effectiveness, safety, and long-term outcomes.

DETAILED DESCRIPTION:
Rationale:

Alopecia areata (AA) is a dermatological disorder characterized by non-scarring hair loss, significantly affecting the quality of life of patients. While some patients experience spontaneous hair regrowth or respond well to localized treatments, patients with moderate-to-severe AA represent a subgroup that requires more extensive systemic therapies for effective management. Currently, the clinical management of moderate-to-severe AA is primarily based on expert opinions. There is a lack of research on systemic treatments for moderate-to-severe AA, comprising only a small number of randomized controlled trials and observational studies. Furthermore, there is a clear absence of long-term, prospective, and comparative data on these therapies. Most conventional systemic treatments for AA are prescribed off-label, underlining the importance of gaining a more comprehensive understanding of their effectiveness and safety.

Therefore, a long-term prospective registry is conducted. This registry will evaluate the real-world utilization of systemic treatments in AA patients, aiming to provide valuable insights into the effectiveness, safety, and long-term outcomes of these therapies. By collecting and analyzing such data, this registry endeavors to contribute to evidence-based clinical management, ultimately improving care for AA patients.

Objective:

The aim is to establish a comprehensive cohort of AA patients receiving systemic treatments, with the primary objective of assessing the short- and long-term effectiveness and safety of various systemic treatments for AA.

Study type:

This is a long-term multicenter prospective, observational, non-interventional registry.

Study population:

All adult AA patients starting systemic treatment, who are willing to provide voluntary informed consent prior to inclusion in the registry and comply with the requirements of the registry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with alopecia areata;
* Starting/using a systemic treatment for alopecia areata;
* Informed consent for registry participation obtained from patient and/or caretaker.

Exclusion Criteria:

* Not sufficiently capable of understanding the Dutch language;
* Not willing to participate.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients with alopecia areata starting/using systemic treatment, who are willing to provide voluntary informed consent prior to inclusion in the registry and comply with the requirements of the registry. All patients will be recruited in the dermatology outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of systemic treatments | A minimum of 10 years from last patient enrolled (every 3-6 months)
  The primary study parameters and endpoints include assessing the short- and long-term effectiveness of various systemic treatments for alopecia areata. Effectiveness ranging from strong improvement to strong deterioration (5 categories).
Safety of systemic treatments | A minimum of 10 years from last patient enrolled (every 3-6 months)
  The primary study parameters and endpoints include assessing the short- and long-term safety of various systemic treatments for alopecia areata. Measured by the number of participants with treatment-related adverse events.

SECONDARY OUTCOMES:
Epidemiological data | Baseline
  Demographics, ethiopathogenesis, co-morbidities, family history, clinical features, treatment history.
Physician Reported - Severity of Alopecia Tool (SALT Score) | A minimum of 10 years from last patient enrolled (every 3-6 months)
  The SALT score measures hair loss on a scale of 0 (no scalp hair loss) to 100 (complete scalp hair loss).
Dermatology Life Quality Index (DLQI, 10 items) | A minimum of 10 years from last patient enrolled (every 3-6 months)
  The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week, scored 0-30.
Alopecia Areata Symptom Impact Scale (AASIS, 13 items) | A minimum of 10 years from last patient enrolled (every 3-6 months)
  The AASIS consists of 13 questions concerning disease-specific patient-reported outcomes measure about symptoms related to alopecia areata and how these symptoms interfere with daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided